CLINICAL TRIAL: NCT06187194
Title: Evaluation of the Efficacy and Safety of an Irreversible Electroporation (IRE) System for Tonsil Reduction for The Treatment of Chronic Symptomatic Tonsillar Hypertrophy
Brief Title: Efficacy and Safety of Irreversible Electroporation for Chronic Symptomatic Tonsillar Hypertrophy Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENTire Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0137
Record Dates: First submitted 2023-09-06; First posted 2024-01-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tonsillar Hypertrophy

STUDY DESIGN:
Intervention Model Description: Irreversible Electroporation (IRE) System for Tonsil Reduction for The Treatment of Chronic Symptomatic Tonsillar Hypertrophy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enlarged tonsil(s) mass will be reduced by ENTire IRE System. (Experimental): The bi-polar IRE System locally applies short, high-voltage (HV) pulses, increasing the permeability of tissue cells, creating non-thermal irreversible electroporation (NTIRE). The energy is transferred via bipolar forceps and causes irreversible cell membrane perforation and apoptosis. This results in tissue reduction within 2-4 weeks after treatment.
  Interventions: Device: IRE System

INTERVENTIONS:
Device: IRE System — Irreversible Electroporation (IRE) System for Tonsil Reduction for The Treatment of Chronic Symptomatic Tonsillar Hypertrophy
  Other Names: ENtire IRE System

SUMMARY:
The purpose of the IRE System is to address the clinical need for reducing the volume of chronic symptomatic hypertrophic tonsil(s) while minimizing side effects and complications. Procedure time will also be reduced. The IRE System is designed to be more comfortable for patients, as it employs a noninvasive procedure using a high voltage pulsed electric field to create irreversible nanopores in the cell membrane, leading to cell death and the reduction of tonsil volume.

DETAILED DESCRIPTION:
The purpose of the IRE System is to address the clinical need for reducing the volume of chronic symptomatic hypertrophic tonsil(s) while minimizing side effects and complications. Procedure time will also be reduced. The IRE System is designed to be more comfortable for patients, as it employs a noninvasive procedure using a high voltage pulsed electric field to create irreversible nanopores in the cell membrane, leading to cell death and the reduction of tonsil volume. On basis of these finding and in view of the known safety profile (refer to Chen et.al ) and efficacy of current technologies, the purpose of the current study is to prospectively determine the efficacy and safety of the IRE System in tonsillar reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years.
* Tonsillar Hypertrophy of grade 2 or higher on the BGST.

Exclusion Criteria:

* Age below 18 years.
* Patients with a pacemaker or similar electro stimulator.
* Patients for whom the anesthesia involves high risk.
* Epilepsy or other condition involving convulsions.
* Inability to give informed consent and to complete self-reported questionnaires.
* Patients with an inability to cooperate for treatment and follow-up.
* Severe heart disease.
* Pregnancy or breastfeeding.
* Significant systemic illness (e.g., cancer, severe autoimmune disease, neurological disease).
* Bleeding diathesis.
* Patients suffering from obesity as indicated by a body mass index (BMI) > 32kg/m2.
* Known or suspected complications for any general or local anesthetic agents and/or any antibiotic medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change of tonsil(s) size in accordance with the Brodsky Grading System for Tonsils (BGST) by at least one grade at 3 months compared to the Baseline. | 3 months popst treatment
  Change of tonsillar hypertrophy by at least one grade and a change in post procedure related pain as compared to literature for other surgical treatment for reducing tonsil tissue mass.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Mary Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No